CLINICAL TRIAL: NCT00938626
Title: Induction of Anti-Myeloma Stem Cell Immunity With Infusions of Autologous Activated T Cells Armed With OKT3 x Rituxan (Anti-CD3 x Anti-CD20) Bispecific Antibody (CD20Bi) (Phase I).
Brief Title: Treated T Cells Followed by a Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Zonder, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000646891; P30CA022453 (NIH); WSU-2008-106
Record Dates: First submitted 2009-07-11; First posted 2009-07-14 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Armed-activated T cells/Immunotherapy (Experimental): At least 1-3 weeks after the second infusion, patients receive high-dose chemotherapy and then undergo autologous peripheral blood stem cell transplantation. Patients then undergo leukapheresis for G-CSF-mobilized autologous T-cells.
  Interventions: Biological: anti-CD3 x anti-CD20 bispecific antibody-armed activated T cells; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: anti-CD3 x anti-CD20 bispecific antibody-armed activated T cells — After completion of induction or salvage chemotherapy, patients receive immunotherapy comprising anti-CD3 x anti-CD20-armed ATC IV weekly for 2 weeks.
Procedure: autologous hematopoietic stem cell transplantation — At least 1-3 weeks after the second infusion, patients receive high-dose chemotherapy and then undergo autologous peripheral blood stem cell transplantation. Patients then undergo leukapheresis for G-CSF-mobilized autologous T-cells.
Procedure: peripheral blood stem cell transplantation — At least 1-3 weeks after the second infusion, patients receive high-dose chemotherapy and then undergo autologous peripheral blood stem cell transplantation.

SUMMARY:
RATIONALE: Giving chemotherapy followed by treated T cells before a stem cell transplant stops the growth of cancer cells by stopping them from dividing or by killing them. After treatment, stem cells are collected from the patient's blood and stored. High-dose chemotherapy is given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This phase I trial is studying the side effects and best way to give treated T cells followed by stem cell transplant in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To test the feasibility and safety of infusing anti-CD3 x anti-CD20 bispecific antibody-armed activated T cells (CD20Bi-AATC) before stem cell mobilization and collection for autologous peripheral blood stem cell transplantation (PBSCT) in patients with multiple myeloma.

Secondary

* To explore functional changes in immune cell populations as a consequence of immunotherapy to test the hypothesis that CD20Bi-AATC can induce anti-clonogenic myeloma precursor cell (CMPC) effect as measured by cytotoxicity; serum cytokine levels; and serum antibody titers to myeloma cells pre-immunotherapy, after immunotherapy, and after high-dose chemotherapy and autologous PBSCT.
* To explore whether the infusion of CD20Bi-AATC reduces the proportion of plasma cells with the CD20+ CMPC phenotype in patients' bone marrow as assessed by multi-color flow cytometry before and after immunotherapy.
* To assess the proportion of bone marrow colony-forming assays before induction or salvage chemotherapy, pre-immunotherapy, and post-immunotherapy to determine whether the infusion grossly affects the bone marrow progenitor populations.
* To explore whether infusions of CD20Bi-AATC induce a B-cell defect causing an immunoglobulin deficiency after autologous PBSCT.
* To measure immunoglobulin deficiency after autologous PBSCT (e.g., quantitative IgG, IgM, and IgA levels and number of circulating T- and B-cell subsets).

OUTLINE: After completion of induction or salvage chemotherapy, patients receive immunotherapy comprising anti-CD3 x anti-CD20-armed ATC IV weekly for 2 weeks. At least 1-3 weeks after the second infusion, patients receive high-dose chemotherapy and then undergo autologous peripheral blood stem cell transplantation. Patients then undergo leukapheresis for G-CSF-mobilized autologous T-cells.

Blood samples are collected periodically to evaluate antibody titers to recall antigens; serum IgG, IgM, and IgA levels; the proportion of circulating B-cells by phenotyping for CD19, CD20, CD22, CD23, CD4, CD8, and CD38; the ability of peripheral blood mononuclear cells to kill multiple myeloma cell lines or the patient's own cryopreserved myeloma cells via cytotoxicity assays and ELISPOT assays; and human anti-mouse antibody responses to murine IgG2a (OKT3). Bone marrow biopsies are also collected to analyze the phenotype of cells (CD20+, CD138-, CD27+, CD22, etc.) via flow cytometry and the proportion of plasma cells via flow cytometry and hematoxylin-and-eosin staining.

After completion of study treatment, patients are followed up for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Candidate for high-dose chemotherapy and autologous stem cell transplantation
* No definite morphologic evidence of myelodysplasia on pretreatment bone marrow

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 or Karnofsky PS 70-100%
* ANC > 500/mm^3
* Platelet count ≥ 75,000/mm^3
* Total bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 3 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL
* LVEF ≥ 45%
* Corrected pulmonary diffusion capacity ≥ 50%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infections or other severe medical problems such as adrenal dysfunction
* No other active malignancy (except for nonmelanoma skin cancer) that requires myelosuppressive chemotherapy or radiotherapy
* No HIV infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* On-chemotherapy induction with thalidomide or lenalidomide with dexamethasone is allowed
* No prior stem cell transplantation
* No more than 2 prior treatment regimens (including the one during which patients undergo leukapheresis for T-cells)
* No more than 4 courses of lenalidomide in combination with other agents or as a single agent over a 1-year period
* No other concurrent immunotherapy, radiotherapy, chemotherapy, or anti-myeloma therapy at the time of the anti-CD3 x anti-CD20-armed ATC infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cell-based toxicities according to NCI CTCAE v3.0 criteria | Up to week 4 after chemotherapy
Ability to mobilize the number of stem cells required for autologous peripheral blood stem cell transplantation (PBSCT) | By day 30 after autologous stem cell transplant (ASCT)

SECONDARY OUTCOMES:
Engraftment of neutrophils | At day 28 after autologous PBSCT
Functional changes in immune cell populations | Prior to immunotherapy (IT), after IT, high dose chemotherapy (HDC)/ autologous stem cell transplant (ASCT) and boost infusion
Assess proportion of erythroid blast-forming unit (BFU)-E, colony forming unit-granulocyte-macrophage (CFU)-GM, CFU-GEMM (granulocyte, erythrocyte, monocyte, megakaryocyte) & erythroid colony forming (CFU-E) | Prior to induction or salvage chemotherapy; Pre & post IT
  To determine whether infusions of CD20 Bi-AATC grossly affected the bone marrow progenitor populations.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Zonder, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States